CLINICAL TRIAL: NCT04812366
Title: Genomic Biomarker-Selected Umbrella Neoadjuvant Study for High Risk Localized Prostate Cancer
Acronym: GUNS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Janssen Inc. (Industry); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Martin Gleave, Principal Investigator/Study Chair, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-03434
Record Dates: First submitted 2021-03-12; First posted 2021-03-23 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Abiraterone Acetate; Prednisone; Docetaxel; niraparib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group 1a (Active Comparator): LHRHa plus apalutamide.
  Interventions: Drug: Apalutamide 60mg Tab
- Group 1b (Active Comparator): LHRHa plus apalutamide plus abiraterone acetate plus prednisone.
  Interventions: Drug: Apalutamide 60mg Tab; Drug: Abiraterone Acetate 250mg; Drug: Prednisone 5mg Tab
- Group 2a (Active Comparator): LHRHa plus abiraterone acetate plus prednisone.
  Interventions: Drug: Abiraterone Acetate 250mg; Drug: Prednisone 5mg Tab
- Group 2b (Active Comparator): LHRHa plus abiraterone acetate plus prednisone plus docetaxel.
  Interventions: Drug: Abiraterone Acetate 250mg; Drug: Prednisone 5mg Tab; Drug: Docetaxel
- Group 3 (Active Comparator): LHRHa plus abiraterone acetate plus prednisone plus niraparib
  Interventions: Drug: Abiraterone Acetate 250mg; Drug: Prednisone 5mg Tab; Drug: Niraparib 100mg Oral Capsule
- Group 4 (Active Comparator): LHRHa plus apalutamide plus atezolizumab
  Interventions: Drug: Apalutamide 60mg Tab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Apalutamide 60mg Tab — 4 tablets by mouth once a day for 24 weeks
  Arms: Group 1a; Group 1b; Group 4
Drug: Abiraterone Acetate 250mg — 4 tablets by mouth on an empty stomach once a day for 16 weeks
  Arms: Group 1b; Group 2a; Group 2b; Group 3
Drug: Prednisone 5mg Tab — 1 tablet by mouth once daily while taking abiraterone acetate
  Arms: Group 1b; Group 2a; Group 2b; Group 3
Drug: Docetaxel — Infusion every 3 weeks for 6 cycles (each cycle has 3 weeks)
  Arms: Group 2b
Drug: Niraparib 100mg Oral Capsule — 3 capsules by mouth once daily for 16 weeks
  Arms: Group 3
Drug: Atezolizumab — 1200mg infusion every 3 weeks for 6 cycles
  Arms: Group 4

SUMMARY:
The objective of this study is to see if providing an appropriate therapy based on the genomic testing of prostate tumour tissue will result in an improved clinical response.

Each participant will be treated with 8 weeks of a luteinizing hormone-releasing hormone agonist (LHRHa) plus apalutamide (APA) while genome sequence characterization is being done. Participants with biopsy specimens deemed unevaluable for genomic testing will remain on LHRHa plus APA for an additional 16 weeks.

Participants with evaluable tissue will be assigned to one of the open-label sub-studies on the basis of genomic profiling results. Within each group, they will be randomized to a specific treatment arm either LHRHa plus APA alone or adding abiraterone acetate and prednisone, docetaxel or niraparib.

The study will evaluate the response rate and outcomes after radical prostatectomy in each arm of the trial.

DETAILED DESCRIPTION:
This is a multi-centre adaptive multi-arm phase II study. Participants are treated with an induction period of at least 8 weeks of LHRH agonist/antagonist (LHRHa) plus apalutamide (APA) while genome sequence characterization is being done.

Genomic sequencing analysis will be performed centrally by Tempus, a CLIA (Clinical Laboratory Improvement Amendments)-certified laboratory. For the DNA gene profiling, formalin-fixed paraffin-embedded (FFPE) prostate cancer and surrounding healthy tissue from diagnostic biopsies will be used for genetic analysis. Copy number profiling will be performed using array Comparative Genomic Hybridisation (aCGH). Targeted sequencing using MiSeq (Illumina) and Ion Proton (Life Technologies) platforms will be performed to identify mutations in a panel of 648 genes.

Based on previous studies, we conservatively expect up to 25% of unevaluable needle biopsy specimens with inadequate/insufficient tumor tissue for genome sequencing. The patients with unevaluable tissue will continue on the master protocol (LHRHa + APA) for an additional 16 weeks followed by radical prostatectomy.

The genomically evaluable patients will be assigned to a specific sub-protocol according to the results of the genomic profile and randomized to a treatment arm within the sub-protocol for 16 weeks, with additional inclusion and exclusion criteria specified in dedicated sub-protocols. Radical prostatectomy will follow sub-protocol treatment.

Sub-protocol 1 - AR axis: No targetable actionable aberration; presence of TMPRSS2-ERG fusion, CHD1 loss or SPOP mutations: (~50% expected prevalence in study population) randomized to:

1. LHRHa + APA for 16 weeks or
2. LHRHa + APA + AAP (Abiraterone Acetate + Prednisone) for 16 weeks

Sub-protocol 2 - Loss of tumour suppressor genes - PTEN, TP53 or TB loss (~40%, bad prognosis) randomized to:

1. LHRHa + AAP for 16 weeks or
2. LHRHa + AAP + docetaxel for 6 cycles

Sub-protocol 3 - DNA damage response alterations (e.g. BRCA1/2, ATM, FANCONI, CDK12) in 6-8% assigned to:

* LHRHa + AAP + PARP (Poly [ADP-ribose] polymerase) inhibitors (niraparib) for 16 weeks

Sub-protocol 4 - Hypermutation, microsatellite instability (MSI), Lynch syndrome or CDK12 in less than 5% assigned to:

a. LHRHa + APA plus PD-L1 inhibitor (atezolizumab) for 16 weeks

ELIGIBILITY:
Inclusion Criteria:

- I. Males ≥ 18 years of age

II. Histologically confirmed adenocarcinoma of the prostate without pathologic evidence of small cell differentiation at the time of initial diagnosis

III. High-risk localized prostate cancer as defined by:

* PSA (prostate specific antigen) >20, any GS or >8 or
* Gleason pattern 4 in 6 or more systematic cores (pattern 4 must be dominant, ≥50% average across 6 or more systematic cores) or
* ≥ 50% Gleason pattern 4 in 3 or more systematic or Magnetic Resonance Imaging (MRI)-targeted cores and PSA ≥ 20 (may include G4+3 or G4+4 but pattern 4 must be dominant, ≥50% average across 3 or more systematic cores) or
* ≥25% Gleason pattern 5 in 3 or more systematic or MRI-targeted cores (may include G4+5, or G3+5, but pattern 5 must be ≥25% average across 3 or more systematic cores).
* Gleason > 8 or greater on minimum of one core either targeted or systematic biopsy and PSA >20
* Participants with oligometastatic (< 3) metastases by PSMA (Prostate-Specific Membrane Antigen) imaging only who are deemed candidates for radical prostatectomy are eligible

IV. Participants must consent to genetic testing at registration and prior to assignment by a central reference laboratory

V. No prior systemic or localized treatment for prostate cancer. Up to 30 days of LHRHa is allowable prior to treatment.

VI. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1 (Appendix II) and a life expectancy of ≥ 3 years

VII. Participants must have adequate end-organ function and all laboratory tests must be performed within 4 weeks prior to registration into master protocol.

VIII. Participant consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrolment in the trial to document their willingness to participate.

Exclusion Criteria:

- I. Received more than 30 days of LHRHa prior to registration and initiation of LHRHa + APA

II. Stage T4 prostate cancer by clinical examination or radiologic evaluation

III. Hypogonadism or severe androgen deficiency as defined by screening serum testosterone more than 50 ng/dL below the normal range for the institution

IV. Participants with serious illnesses or medical conditions which could cause unacceptable safety risks or would not permit the participant to be managed according to the protocol. This includes but is not limited to:

* Active infection or chronic liver disease requiring systemic therapy;
* Active or known human immunodeficiency virus (HIV) with detectable viral load;
* Uncontrolled or recent clinically significant cardiac disease, including: angina pectoris, symptomatic pericarditis, coronary artery bypass grafting, coronary angioplasty, or stenting, or myocardial infarction in the previous 12 months; history of documented congestive heart failure (New York Heart Association functional classification III-IV) or cardiomyopathy; history of any cardiac arrhythmias, e.g. ventricular, supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months;
* Participants with uncontrolled hypertension

V. Participants who are unable to swallow oral medication and/or have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)

VI. Participants with a history of hypersensitivity to any of the study drugs or any excipient

VII. Participants with a history of non-compliance to medical regimen

VIII. Severe concurrent disease, infection, or co-morbidity that, in the judgement of the Investigator, would make the participant inappropriate for enrollment or prostatectomy

IX. Prior androgen deprivation, chemotherapy, surgery, or radiation for prostate cancer

X. Receiving concurrent androgens, estrogens, or pregestational agents, or prior exposure to any of these agents within 6 months prior to randomization

XI. M1 by conventional imaging (CT, bone scan)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a prostate cancer study
Enrollment: 315 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete Pathologic Response (pCR) | 6 years
  Pathological Minimal Residual Disease (pMRD): pathological minimal residual disease (pMRD) is defined as residual tumour 5mm or less.
Pathological Minimal Residual Disease (pMRD) | 6 years
  Pathological minimal residual disease is defined as residual tumour 5 mm or less.

SECONDARY OUTCOMES:
Pain level assessment | 6 years
  The Brief Pain Inventory-Short Form (BPI-SF) is a 9-item, self administered questionnaire which evaluates the severity of a participant's level of pain and impact on daily functioning. This questionnaire will be administered at screening, prior to receiving master protocol therapy (0 weeks), the end of receiving therapy (8 weeks), as well as the End of Treatment (EoT) visit.
Generic Quality of Life (QoL) | 6 years
  The EQ-5D-5L is a widely used instrument developed in Europe to evaluate the generic quality of life. The EQ-5D-5L has two components: the EQ-5D descriptive system and the EQ visual analogue scale. This questionnaire will be administered at screening, prior to receiving master protocol therapy (0 weeks), the end of receiving therapy (8 weeks) as well as at the EoT visit.
Quality of Life-Prostate Cancer Patients | 6 years
  This will be measured using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire. The FACT-P is a multidimensional, self-report QoL instrument specifically designed for use with patients who have prostate cancer. This questionnaire will be administered at screening, prior to receiving master protocol therapy (0 weeks), the end of receiving therapy (8 weeks) as well as at the EoT visit.

CONTACTS AND LOCATIONS:
Overall Officials: Martin E Gleave, MD, Study Chair — University of British Columbia
Locations (9):
- United States (5):
  - University of California Davis, Sacramento, California
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - U.T. MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Canada (4):
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Research Institute (OHRI), Ottawa, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No